CLINICAL TRIAL: NCT05453162
Title: Circadian Influence on Fear Extinction Resulting From Prolonged Exposure Therapy for PTSD
Brief Title: Circadian Influence on Prolonged Exposure Therapy for PTSD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: VA Boston Healthcare System (U.S. Federal Agency); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Edward F. Pace-Schott, Assistant Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021p003356; R21MH128619 (NIH)
Record Dates: First submitted 2022-06-29; First posted 2022-07-12 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: PTSD
Keywords: PTSD; Circadian; Exposure Therapy; Sleep; Cortisol
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants (52 total) will be randomized, 26 to each of 2 arms one of which has 8 weekly PE sessions in early morning (between 07:00-10:00) and the other 8 sessions PE at 16:00 or later. Homework exposures will occur at the same time of day as PE. Primary outcomes measured at beginning, middle and end of treatment will be psychophysiological reactivity to trauma recall (mechanistic outcome) and CAPS-5 (clinical outcome). Secondary mechanistic outcome is peak SUDS during PE and clinical is PCL-5 measured at each PE session. Endogenous salivary cortisol levels will be tested as a mechanism of circadian effect. Data will be analyzed using multilevel, mixed-effects models.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Therapists will be unaware of study hypotheses. therapy supervisor and assessors will be unaware of hypothesis and participants' treatment arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early morning PE (Experimental): 26 participants randomized to 10 weekly PE sessions in early morning (between 07:00-10:00) with homework exposures occurring occur at this same time of day.
  Interventions: Behavioral: Prolonged Exposure Therapy for Posttraumatic Stress Disorder
- Late afternoon PE (Experimental): 26 participants randomized to 10 weekly PE sessions in late afternoon (16:00 or later) with homework exposures occurring occur at this same time of day.
  Interventions: Behavioral: Prolonged Exposure Therapy for Posttraumatic Stress Disorder

INTERVENTIONS:
Behavioral: Prolonged Exposure Therapy for Posttraumatic Stress Disorder — Manualized procedures deliver ten 90-minute sessions targeted to occur weekly and administered via tele-health with the same study therapist. Session 1 will focus on psychoeducation. Session 2 involves construction of the in vivo exposure hierarchy. Sessions 3-10 focus on in-session imaginal exposures to the worst trauma memory for 45-60 min followed by 15-20 min of processing the imaginal exposure. For homework, participants will be instructed to confront situations on their hierarchy on a daily basis using recording of their imaginal exposure. Subjective Units of Distress (SUDS) ratings will be taken throughout imaginal exposure exercises.

SUMMARY:
Proposed research will examine time-of-day effects on trauma-related fear extinction using Prolonged Exposure Therapy (PE) telemedicine for Posttraumatic Stress Disorder (PTSD) in the National Center for PTSD (NCPTSD). The primary mechanistic outcome measure will be change in psychophysiological reactivity to script-driven imagery (SDI-PR) measured, in person, at pre-treatment, after 5 PE sessions (mid-treatment), and after all 10 PE sessions (post-treatment). A secondary mechanistic outcome will be session-to-session reduction in peak subjective units of distress (SUDS) ratings to imaginal exposures. The primary clinical outcome will be change in Clinican Administered PTSD Scale (CAPS-5) severity score; a secondary clinical outcome will be session-to-session reduction in self-reported PTSD symptoms using the PTSD checklist (PCL-5). Participants meeting inclusion criteria (described below) will be randomized to either PE sessions that begin from 07:00 to a time no later than 2 hours past a participant's customary rise time, or to the last treatment session of the day beginning at 16:00 or later (26 per arm). Participants will complete daily at-home imaginal-exposure homework within the same time frame as their PE sessions are scheduled, i.e., within 2 hours of awakening for morning (AM) group and between 16:00 and 2 hours before bedtime for late afternoon (PM) group.

DETAILED DESCRIPTION:
Proposed research will examine time-of-day effects on trauma-related fear extinction using PE therapy for PTSD in the National Center for PTSD (NCPTSD). The primary mechanistic outcome measure will be change in SDI-PR; a secondary mechanistic outcome will be session-to-session reduction in peak SUDS ratings to imaginal exposures. The primary clinical outcome will be change in CAPS-5 severity score; a secondary clinical outcome will be session-to-session reduction in self-reported PTSD symptoms (PCL-5). Participants meeting inclusion criteria (described below) will be randomized to either PE sessions that begin from 07:00 to a time no later than 2 hours past a participant's customary rise time, or to the last treatment session of the day beginning at 16:00 or later. Participants will complete daily at-home imaginal-exposure homework within the same time frame as their PE sessions are scheduled (i.e., within 2 hours of awakening for morning group and between 16:00 and 2 hours before bedtime for late afternoon group). The assessment schedule will be identical for all participants. Participants who meet study inclusion criteria at screening will first begin a 7-day, pre-study sleep-monitoring period with wrist actigraphy, sleep diaries and completion of a diurnal profile of salivary cortisol levels. Trauma-related fear will be assessed using the standard SDI procedures detailed below at pre-treatment, after 5 PE sessions (mid-treatment), and after all 10 PE sessions (post-treatment). The CAPS-5 will be administered at these same times. PCL-5 measurements will be obtained at each treatment session and SUDs will be obtained during all treatment sessions that include imaginal exposure (sessions 3-8). All SDI sessions will be carried out at a standardized time of day in the late-afternoon (15:00-17:00). PE treatment will be administered at a targeted rate of once per week. At each PE and assessment session, pre-session saliva samples will be obtained for cortisol measurement and normalized using the diurnal profile of cortisol obtained during the sleep-assessment week. Participants will wear the wrist actigraph and complete sleep diaries throughout PE. The diurnal cortisol profile will be repeated at the post-treatment assessment.

ELIGIBILITY:
Inclusion Criteria:

1. a diagnosis of PTSD as defined by DSM-5, with a minimum CAPS severity score of 26, a minimum PCL-5 score of 31, or a score of 2 or above on CAPS-5 Item B2 (concerning distressing dreams)
2. interest in starting a course of PE
3. availability for appointments at that will either begin from 07:00 to a time no longer than 2 hours past their customary rise time, or to the last treatment session of the day beginning at 16:00 or later
4. Age range of 18-70
5. A Morningness-Eveningness Questionnaire (MEQ) score above 25.
6. Non-exclusionary psychotropic medications must have been stable for 3 weeks prior to Screening/Assessment with intention to remain stable throughout participation.

Exclusion Criteria:

1. current or past history of bipolar I disorder, schizophrenic or other psychotic disorders,
2. current organic brain disorder including moderate to severe traumatic brain injury
3. factitious disorder or malingering
4. pregnant or planning to become pregnant in the next four months at time of screening [if a participant does become pregnant during study procedures, the situation will be reviewed on a case-by-case basis and the participant's wishes will be considered in deciding whether the participant will continue with the study or withdraw.]
5. current moderate or severe substance use disorder with symptoms present within the past three months
6. diagnosed moderate to severe sleep apnea, narcolepsy, periodic limb movement, or restless legs syndrome that result in daytime sleepiness indicated by Epworth Sleepiness Scale (ESS) above 10
7. active risk of harm to self or others
8. evidence of clinically significant hepatic or renal disease or any other acute or unstable medical condition that might interfere with safe conduct of the study
9. current participation in trauma-focused cognitive-behavioral therapy (e.g., Cognitive Processing Therapy, Written Exposure Therapy, Eye Movement Desensitization and Reprocessing Therapy)
10. prior treatment with an adequate dose of PE (i.e., 8 or more sessions) to the traumatic event that would be the index trauma for treatment in the study
11. having no memory of their traumatic event
12. daily use of benzodiazepines
13. methadone or suboxone maintenance therapy for past opioid addiction
14. diagnosis of Cushing's disease, Addison's disease or use of medications that target cortisol directly such as those used to treat Cushing's disease [ketoconazole, mitotane (Lysodren), metyrapone (Metopirone), and Mifepristone (Korlym, Mifeprex)], those used to treat Addison's disease [Hydrocortisone (Cortef), prednisone or methylprednisolone], as well as cortisone or dexamethasone.
15. persons who would habitually awaken so early that more than 2 h would elapse before a morning PE session could occur; or those who engage in habitual shiftwork or transmeridian travel

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Psychophysiological reactivity to script-driven imagery (SDI-PR): Primary Mechanistic Outcome | Between days -7 to -1, Baseline
  This primary mechanistic outcome is a unitary discriminant canonical variable measuring psychophysiological reactivity while listening to personalized recorded scripts describing an index trauma.
Psychophysiological reactivity to script-driven imagery (SDI-PR): Primary Mechanistic Outcome | Between days 29-34, mid-treatment
  This primary mechanistic outcome is a unitary discriminant canonical variable measuring psychophysiological reactivity while listening to personalized recorded scripts describing an index trauma.
Psychophysiological reactivity to script-driven imagery (SDI-PR: )Primary Mechanistic Outcome | Between days 64-71, post-treatment
  This primary mechanistic outcome is a unitary discriminant canonical variable measuring psychophysiological reactivity while listening to personalized recorded scripts describing an index trauma.
Clinician-Administered PTSD scale for Diagnostic and Statistical Manual of Mental Disorders (DSM), Fifth Edition (CAPS-5): Primary Clinical Outcome | Between days -7 to -1, Baseline
  This primary clinical outcome is the gold standard clinical interview for assessing PTSD severity. In CAPS-5, each of the 20 symptoms of PTSD is rated on a 5-point severity scale ranging from 0 (absent) to 4 (extreme). Total scores range from 0 to 80.
CAPS-5: Primary Clinical Outcome | Between days 29-34, mid-treatment
  This primary clinical outcome is the gold standard clinical interview for assessing PTSD severity. In CAPS-5, each of the 20 symptoms of PTSD is rated on a 5-point severity scale ranging from 0 (absent) to 4 (extreme). Total scores range from 0 to 80.
CAPS-5: Primary Clinical Outcome | Between days 64-71, post-treatment
  This primary clinical outcome is the gold standard clinical interview for assessing PTSD severity. In CAPS-5, each of the 20 symptoms of PTSD is rated on a 5-point severity scale ranging from 0 (absent) to 4 (extreme). Total scores range from 0 to 80.

SECONDARY OUTCOMES:
Subjective Units of Distress (SUDS): Secondary Mechanistic Outcome | Day 14 Peak SUDS during PE therapy session 3
  A rating scale from 0 to 100 where zero represents no distress at all and 100 represents very extreme distress, fear, or anxiety. SUDS ratings are subjective and different individuals may rate the same situation differently. An individual anchors their own ratings with personal recollection of situations considered "No Distress" to "Moderate" to "Extreme Distress".
SUDS: Secondary Mechanistic Outcome | Day 21 Peak SUDS during PE therapy session 4
  A rating scale from 0 to 100 where zero represents no distress at all and 100 represents very extreme distress, fear, or anxiety. SUDS ratings are subjective and different individuals may rate the same situation differently. An individual anchors their own ratings with personal recollection of situations considered "No Distress" to "Moderate" to "Extreme Distress".
SUDS: Secondary Mechanistic Outcome | Day 28 Peak SUDS during PE therapy session 5
  A rating scale from 0 to 100 where zero represents no distress at all and 100 represents very extreme distress, fear, or anxiety. SUDS ratings are subjective and different individuals may rate the same situation differently. An individual anchors their own ratings with personal recollection of situations considered "No Distress" to "Moderate" to "Extreme Distress".
SUDS: Secondary Mechanistic Outcome | Day 35 Peak SUDS during PE therapy session 6
  A rating scale from 0 to 100 where zero represents no distress at all and 100 represents very extreme distress, fear, or anxiety. SUDS ratings are subjective and different individuals may rate the same situation differently. An individual anchors their own ratings with personal recollection of situations considered "No Distress" to "Moderate" to "Extreme Distress".
SUDS: Secondary Mechanistic Outcome | Day 42 Peak SUDS during PE therapy session 7
  A rating scale from 0 to 100 where zero represents no distress at all and 100 represents very extreme distress, fear, or anxiety. SUDS ratings are subjective and different individuals may rate the same situation differently. An individual anchors their own ratings with personal recollection of situations considered "No Distress" to "Moderate" to "Extreme Distress".
SUDS: Secondary Mechanistic Outcome | Day 49 Peak SUDS during PE therapy session 8
  A rating scale from 0 to 100 where zero represents no distress at all and 100 represents very extreme distress, fear, or anxiety. SUDS ratings are subjective and different individuals may rate the same situation differently. An individual anchors their own ratings with personal recollection of situations considered "No Distress" to "Moderate" to "Extreme Distress".
SUDS: Secondary Mechanistic Outcome | Day 56 Peak SUDS during PE therapy session 9
  A rating scale from 0 to 100 where zero represents no distress at all and 100 represents very extreme distress, fear, or anxiety. SUDS ratings are subjective and different individuals may rate the same situation differently. An individual anchors their own ratings with personal recollection of situations considered "No Distress" to "Moderate" to "Extreme Distress".
SUDS: Secondary Mechanistic Outcome | Day 63 Peak SUDS during PE therapy session 10
  A rating scale from 0 to 100 where zero represents no distress at all and 100 represents very extreme distress, fear, or anxiety. SUDS ratings are subjective and different individuals may rate the same situation differently. An individual anchors their own ratings with personal recollection of situations considered "No Distress" to "Moderate" to "Extreme Distress".
PCL-5: PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM), Fifth Edition: Secondary Clinical Outcome | Day 0 PCL-5 score at PE therapy session 1
  Self-ratings of how much one is bothered by each of the 20 symptoms of PTSD on a 5-point severity scale ranging from 0 (Not at all) to 4 (extremely).
PCL-5: Secondary Clinical Outcome | Day 7 PCL-5 score at PE therapy session 2
  Self-ratings of how much one is bothered by each of the 20 symptoms of PTSD on a 5-point severity scale ranging from 0 (Not at all) to 4 (extremely).
PCL-5: Secondary Clinical Outcome | Day 14 PCL-5 score at PE therapy session 3
  Self-ratings of how much one is bothered by each of the 20 symptoms of PTSD on a 5-point severity scale ranging from 0 (Not at all) to 4 (extremely).
PCL-5: Secondary Clinical Outcome | Day 21 PCL-5 score at PE therapy session 4
  Self-ratings of how much one is bothered by each of the 20 symptoms of PTSD on a 5-point severity scale ranging from 0 (Not at all) to 4 (extremely).
PCL-5: Secondary Clinical Outcome | Day 28 PCL-5 score at PE therapy session 5
  Self-ratings of how much one is bothered by each of the 20 symptoms of PTSD on a 5-point severity scale ranging from 0 (Not at all) to 4 (extremely).
PCL-5: Secondary Clinical Outcome | Day 35 PCL-5 score at PE therapy session 6
  Self-ratings of how much one is bothered by each of the 20 symptoms of PTSD on a 5-point severity scale ranging from 0 (Not at all) to 4 (extremely).
PCL-5: Secondary Clinical Outcome | Day 42 PCL-5 score at PE therapy session 7
  Self-ratings of how much one is bothered by each of the 20 symptoms of PTSD on a 5-point severity scale ranging from 0 (Not at all) to 4 (extremely).
PCL-5: Secondary Clinical Outcome | Day 49 PCL-5 score at PE therapy session 8
  Self-ratings of how much one is bothered by each of the 20 symptoms of PTSD on a 5-point severity scale ranging from 0 (Not at all) to 4 (extremely).
PCL-5: Secondary Clinical Outcome | Day 56 PCL-5 score at PE therapy session 9
  Self-ratings of how much one is bothered by each of the 20 symptoms of PTSD on a 5-point severity scale ranging from 0 (Not at all) to 4 (extremely).
PCL-5: Secondary Clinical Outcome | Day 63 PCL-5 score at PE therapy session 10
  Self-ratings of how much one is bothered by each of the 20 symptoms of PTSD on a 5-point severity scale ranging from 0 (Not at all) to 4 (extremely).

OTHER OUTCOMES:
Salivary cortisol | Between days -7 to -1, baseline
  Concentration in saliva sample obtained by passive drool and analyzed by enzyme immunoassay
Salivary cortisol | Day 0, therapy session 1
  Concentration in saliva sample obtained by passive drool and analyzed by enzyme immunoassay
Salivary cortisol | Day 7, therapy session 2
  Concentration in saliva sample obtained by passive drool and analyzed by enzyme immunoassay
Salivary cortisol | Day 14, therapy session 3
  Concentration in saliva sample obtained by passive drool and analyzed by enzyme immunoassay
Salivary cortisol | Day 21, therapy session 4
  Concentration in saliva sample obtained by passive drool and analyzed by enzyme immunoassay
Salivary cortisol | Day 28, therapy session 5
  Concentration in saliva sample obtained by passive drool and analyzed by enzyme immunoassay
Salivary cortisol | Between days 29-34, mid-treatment assessment
  Concentration in saliva sample obtained by passive drool and analyzed by enzyme immunoassay
Salivary cortisol | Day 35, therapy session 6
  Concentration in saliva sample obtained by passive drool and analyzed by enzyme immunoassay
Salivary cortisol | Day 42, therapy session 7
  Concentration in saliva sample obtained by passive drool and analyzed by enzyme immunoassay
Salivary cortisol | Day 49, therapy session 8
  Concentration in saliva sample obtained by passive drool and analyzed by enzyme immunoassay
Salivary cortisol | Day 56, therapy session 9
  Concentration in saliva sample obtained by passive drool and analyzed by enzyme immunoassay
Salivary cortisol | Day 63, therapy session 10
  Concentration in saliva sample obtained by passive drool and analyzed by enzyme immunoassay
Salivary cortisol | Between days 64-71, post-treatment
  Concentration in saliva sample obtained by passive drool and analyzed by enzyme immunoassay

CONTACTS AND LOCATIONS:
Overall Officials: Edward F Pace-Schott, PhD, Principal Investigator — Massachusetts General Hospital; Suzanne L Pineles, PhD, Principal Investigator — VA Boston Health System, Boston University
Locations (1):
- VA Boston Healthcare System, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share data every January 15 and July 15 with the NIMH Data Archives (NDA) under a NIMH Data Repositories Data Submission Agreement between NIMH and VA Boston Health System (VABHS). Data sharing is required for all NIMH-funded research projects. The NDA DSA will be approved by the VABHS IRB. Each participant will be assigned Global Unique ID (GUID) and data shared will contain no identifiable information. Shared data will include scored psychophysiological, self-report instruments, cortisol, actigraphy, and fully de-identified demographic data.
Supporting Information: Study Protocol
Time Frame: Study data will become available following the end of the study and the publication of results.
Access Criteria: Investigators can apply to the NIMH Data Archive (NDA) for permission to use these data.
URL: https://nda.nih.gov

REFERENCES:
- [Background] Pace-Schott EF, Spencer RM, Vijayakumar S, Ahmed NA, Verga PW, Orr SP, Pitman RK, Milad MR. Extinction of conditioned fear is better learned and recalled in the morning than in the evening. J Psychiatr Res. 2013 Nov;47(11):1776-84. doi: 10.1016/j.jpsychires.2013.07.027. Epub 2013 Aug 28. PMID 23992769
- [Background] Pace-Schott EF, Germain A, Milad MR. Effects of sleep on memory for conditioned fear and fear extinction. Psychol Bull. 2015 Jul;141(4):835-57. doi: 10.1037/bul0000014. Epub 2015 Apr 20. PMID 25894546
- [Background] Meuret AE, Rosenfield D, Bhaskara L, Auchus R, Liberzon I, Ritz T, Abelson JL. Timing matters: Endogenous cortisol mediates benefits from early-day psychotherapy. Psychoneuroendocrinology. 2016 Dec;74:197-202. doi: 10.1016/j.psyneuen.2016.09.008. Epub 2016 Sep 15. PMID 27664810
- [Background] Pace-Schott EF, Germain A, Milad MR. Sleep and REM sleep disturbance in the pathophysiology of PTSD: the role of extinction memory. Biol Mood Anxiety Disord. 2015 May 29;5:3. doi: 10.1186/s13587-015-0018-9. eCollection 2015. PMID 26034578
- [Background] Meuret AE, Trueba AF, Abelson JL, Liberzon I, Auchus R, Bhaskara L, Ritz T, Rosenfield D. High cortisol awakening response and cortisol levels moderate exposure-based psychotherapy success. Psychoneuroendocrinology. 2015 Jan;51:331-40. doi: 10.1016/j.psyneuen.2014.10.008. Epub 2014 Oct 16. PMID 25462905
- [Background] Brueckner AH, Lass-Hennemann J, Wilhelm FH, Ferreira de Sa DS, Michael T. Cortisol administration after extinction in a fear-conditioning paradigm with traumatic film clips prevents return of fear. Transl Psychiatry. 2019 Apr 8;9(1):128. doi: 10.1038/s41398-019-0455-0. PMID 30962423